CLINICAL TRIAL: NCT02282332
Title: The Impact of Ticagrelor on Coronary Atherosclerotic Lipid Pool and Inflammation Assessed by Near-Infrared Spectroscopy
Brief Title: NIRS Ticagrelor Evaluation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AZ_ISSBRIL0304
Record Dates: First submitted 2014-10-15; First posted 2014-11-04 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patiens Discharged on Ticagrelor (Experimental): Patients to be discharged on ticagrlore regiment of 90mg twice a day for 6 months.
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor

SUMMARY:
The Impact of Ticagrelor on Coronary Atherosclerotic Lipid Pool and Inflammation Assessed by Near-Infrared Spectroscopy study will evaluate whether ticagrelor leads to a 20% reduction in the LCBI with NIRS/IVUS suggesting coronary plaque stabilization and reduced inflammation in patients already on long-term statin therapy undergoing non-urgent PCI. It is hypothesized that the treatment with ticagrelor following PCI will lead to a significant 20% reduction in the lipid pool as measured by NIRS/IVUS at follow-up when compared with baseline imaging, suggesting a reduction in inflammation and stabilization of the lipid core in atherosclerotic lesions not treated during the index procedure.

DETAILED DESCRIPTION:
Single-Center, open-label study of the effect of ticagrelor on the reduction in the lipid pool in 30 patients with multi-vessel CAD 2 Treatment periods over 6 months, with 2 additional follow-up phone calls at 1 and 3 months.

Non-urgent PCI requiring stent placement and evaluation by NIRS/IVUS at baseline and 6 month follow up A second concomitant coronary lesion with diameter stenosis greater than 50% will also be imaged using NIRS/IVUS.

Patients will be discharged on a ticagrelor regiment of 90 mg twice a day for the 6 month study.

Blood samples will be drawn at baseline prior to ticagrelor being administered and again at follow up.

Inclusion Criteria:

* Female (post menopausal or surgically sterile) and/or male aged 18 years or older
* Multi-vessel coronary artery disease
* Statin therapy for minimum of 6 weeks prior to enrollment in the study with no plan for further adjustment
* Non-emergent PCI for ACS with stent placement requiring dual-antiplatelet therapy
* Ability to safely perform NIRS/IVUS for a concomitant non-culprit lesion with diameter stenosis ≥ 50% that was not treated with PCI
* Willing and able to sign informed consent and participate in follow-up

Exclusion Criteria:

* Thienopyridine or ticagrelor use in the last month
* Need for coronary artery bypass surgery or other surgeries during the follow-up period
* Documented medication non-compliance
* Chronic inflammatory disorder or treatment with anti-inflammatory or immunosuppressive drugs
* Prior or current malignancy within the last 5 years
* Concomitant severe illness or reduced life expectancy that will prevent follow-up cardiac catheterization
* Active infection
* Pregnant or lactating women
* End-stage renal disease
* History of intracranial hemorrhage
* Active pathological bleeding
* Known sever hepatic impairment
* Known hypersensitivity to ticagrelor

Study Procedures:

After consent is obtained non-urgent PCI requiring stent placement and evaluation by NIRS/IVUS at baseline is performed and once again at 6 month follow up. A second concomitant coronary lesion with diameter stenosis greater than 50% will also be imaged using NIRS/IVUS. Patients will be discharged on a ticagrelor regiment of 90 mg twice a day for the 6 month study.Blood samples will be drawn at baseline prior to ticagrelor being administered and again at follow up. There will be 1 month phone follow up, 3 month phone follow up and a 6 month clinical follow up that includes collecting blood, repeat catheterization, and repeat NIRS/IVUS procedure.

ELIGIBILITY:
Inclusion Criteria:

* • Female (post menopausal or surgically sterile) and/or male aged 18 years or older

  * Multi-vessel coronary artery disease CAD
  * Statin therapy for minimum of 6 weeks prior to enrollment in the study with no plan for further adjustment
  * Non-emergent PCI for ACS with stent placement requiring dual-antiplatelet therapy
  * Ability to safely perform NIRS/IVUS for a concomitant non-culprit lesion with diameter stenosis ≥50% that was not treated with PCI
  * Willing and able to sign informed consent and participate in follow-up

Exclusion Criteria:

* Thienopyridine or ticagrelor use in the last month
* Need for coronary artery bypass surgery or other surgeries during the follow-up period
* Documented medication non-compliance
* Chronic inflammatory disorder or treatment with anti-inflammatory or immunosuppressive drugs
* Prior or current malignancy within the last 5 years
* Concomitant severe illness or reduced life expectancy that will prevent follow-up cardiac catheterization
* Active infection
* Pregnant or lactating women
* End-stage renal disease
* History of intracranial hemorrhage
* Active pathological bleeding
* Known severe hepatic impairment
* Known hypersensitivity to ticagrelor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Patiens Discharged on Ticagrelor: Patients to be discharged on ticagrlore regiment of 90mg twice a day for 6 months.
  Ticagrelor
Period: Overall Study
Arm/Group | Patiens Discharged on Ticagrelor
Started | 0 (The PI has left the institution and no results data is available. Efforts were made to contact the PI/study team members, as well as to review data on shared drives, IRB historical records and published resources, but were unsuccessful. No study data are available)
Completed | 0 (The PI has left the institution and no results data is available. Efforts were made to contact the PI/study team members, as well as to review data on shared drives, IRB historical records and published resources, but were unsuccessful. No study data are available)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The PI has left the institution and no results data is available. Efforts were made to contact the PI/study team members, as well as to review data on shared drives, IRB historical records and published resources, but were unsuccessful. No study data are available
Arm/Group | Patiens Discharged on Ticagrelor
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Lipid Pool to Follow up as Assessed by NIRS/IVUS With Treatment of Ticagrelor
Description: Treatment with ticagrelor following PCI will lead to significant 20% reduction in the LCBI as assessed at follow up by NIRS/IVUS when compared with baseline imaging data of the reference vessel, suggesting a reduction in inflammation and stabilization of the lipid core in atherosclerotic lesions not treated during the index procedure.
Time Frame: 6 months
Population: as for baseline characteristics
Arm/Group | Patiens Discharged on Ticagrelor
Number analyzed (Participants) | 0

2. Secondary Outcome: Change From Baseline Inflammatory Markers to Follow up With Treatment of Ticagrelor
Description: We expect to see a significant reduction of inflammatory markers of Hs-CRP, MCP-1, IL-1, IL-6, IL-18, and TNF- α as well as an increase in IL-10, a cytokine associated with a reduction in inflammation, following therapy with ticagrelor when compared with baseline values. This is expected as inflammatory markers should be lower in stable coronary artery disease compared with patients presenting with ACS. While there is no control group in the proposed study, it will be important to assess whether changes in established biomarkers associated with inflammation correlate with changes in LCBI. While ticagrelor was not shown to reduce inflammatory biomarkers to a greater degree than clopidogrel, it will be important to assess whether the reduction in LCBI is independent of or associated with reductions in inflammatory markers or platelet reactivity.
Time Frame: 6 months
Population: as for baseline characteristics
Arm/Group | Patiens Discharged on Ticagrelor
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The PI has left the institution and no results data is available. Efforts were made to contact the PI/study team members, as well as to review data on shared drives, IRB historical records and published resources, but were unsuccessful. No study data are available
Arm/Group | Patiens Discharged on Ticagrelor
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No